CLINICAL TRIAL: NCT00191334
Title: Phase II Study of Gemcitabine Plus Cisplatin as First-Line Therapy in Patients With Epithelial Ovarian Cancer
Brief Title: Gemcitabine in Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9340; B9E-MW-S368
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Results first posted 2009-03-27 (Estimated); Last update posted 2009-03-27 (Estimated); Status verified 2009-02

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Drug: gemcitabine; Drug: cisplatin

INTERVENTIONS:
Drug: gemcitabine — 1250 mg/m2, intravenous (IV) day 1 and day 8, every 21 days x 6 cycles or disease progression or unacceptable toxicity
  Other Names: LY188011; Gemzar
Drug: cisplatin — 75 mg/m2, intravenous (IV), every 21 days x 6 cycles or disease progression or unacceptable toxicity

SUMMARY:
The primary endpoint of this study is to assess the objective tumor response rate in patients with advanced epithelial ovarian cancer receiving combination of Gemcitabine at a dose 1250 mg/m2 (Day 1 and 8) with Cisplatin 75 mg/m2 (Day 1) as first-line treatment

ELIGIBILITY:
Inclusion Criteria:

* ECOG = 0-2
* Operated patients
* disease stage III-IV

Exclusion Criteria:

* No prior chemotherapy or radiation therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2004-12; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (5):
- Russia (5):
  - For additional information regarding investigative sites for thsi trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Irkutsk
  - For additional information regarding investigative sites for thsi trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ivanovo
  - For additional information regarding investigative sites for thsi trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Moscow
  - For additional information regarding investigative sites for thsi trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Petersburg
  - For additional information regarding investigative sites for thsi trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Stavropol

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Gemcitabine + Cisplatin: Gemcitabine: 1250 mg/m2, intravenous (IV) day 1 and day 8, every 21 days x 6 cycles or disease progression or unacceptable toxicity.
  Cisplatin: 75 mg/m2, intravenous (IV), every 21 days x 6 cycles or disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Gemcitabine + Cisplatin
Started | 50
Completed | 33
Not Completed | 17
Not completed — Adverse Event | 4
Not completed — Disease Progression or Relapse | 8
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Arm/Group | Gemcitabine + Cisplatin
Number analyzed (Participants) | 50
Age Continuous [Mean (Standard Deviation); unit: years] | 54.9 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50
  Male | 0
Region of Enrollment [Number; unit: participants]
  Russian Federation | 50
Disease Stage [Number; unit: participants]
  Stage I - Tumor Limited to Ovaries | 0
  Stage II - Pelvic Extension and/or Implants | 0
  Stage IIIa - Microscopic Peritoneal Metastasis | 1
  Stage IIIb - Macroscopic Peritoneal Metastasis | 3
  Stage IIIc - Peritoneal Metastasis More Than 2 cm | 21
  Stage IV - Distant Metastases | 25
Eastern Cooperative Oncology Group Performance Status Score [Number; unit: participants]
  0 - Fully Active | 28
  1 - Ambulatory, Restricted Strenuous Activity | 20
  2 - Ambulatory, No Work Activities | 2
  3 - Partially Confined to Bed, Limited Self Care | 0
  4 - Completely Disabled | 0
Postoperational Pathomorphological Diagnosis [Number; unit: participants]
  Serous Cystadenocarcinoma | 37
  Mucinosa Cystadenocarcinoma | 3
  Endometrioid Carcinoma | 4
  Other | 6
Race/Ethnicity [Number; unit: participants]
  Caucasian | 49
  Other | 1
State of Patient Relative to Menopause [Number; unit: participants]
  Fertile Period | 4
  Post-Menopause | 46
Time from Initial Diagnosis to Study Entry [Mean (Standard Deviation); unit: days] | 14.0 (10.3)

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Tumor Response
Description: Best response recorded from the start of treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the treatment started).
Time Frame: every other 21 day cycle (6-8 cycles), every 3 months during long-term follow-up
Measure: Number; unit: participants
Arm/Group | Gemcitabine + Cisplatin
Number analyzed (Participants) | 50
participants
  Complete Response | 6
  Partial Response | 25
  Stable Disease | 10
  Progressive Disease | 5
  Not Assessed | 4

2. Secondary Outcome: Duration of Response
Description: The duration of a complete response (CR) or partial response (PR) was defined as the time from first objective status assessment of CR or PR to the first time of progression or death as a result of any cause.
Time Frame: every other 21 day cycle (6-8 cycles) and every 3 months during long-term follow-up
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Gemcitabine + Cisplatin
Number analyzed (Participants) | 50
weeks | 37.0 [31.1 to 51.1]

3. Secondary Outcome: Time to Progressive Disease
Description: Defined as the time from study enrollment to the first date of disease progression. Time to disease progression was censored at the date of death if death was due to other cause.
Time Frame: every other 21 day cycle (6-8 cycles) and every 3 months during long-term follow-up
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Gemcitabine + Cisplatin
Number analyzed (Participants) | 50
weeks | 45.1 [37.9 to 56.9]

4. Secondary Outcome: Time to Treatment Failure
Description: Defined as the time from study enrollment to the first observation of disease progression, death as a result of any cause, or early discontinuation of treatment. Time to treatment failure was censored at the date of the last follow-up visit for patients who did not discontinue early, who were still alive, and who have not progressed.
Time Frame: every other 21 day cycle (6-8 cycles) and every 3 months during long-term follow-up
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Gemcitabine + Cisplatin
Number analyzed (Participants) | 50
weeks | 38.4 [29.1 to 48.3]

5. Secondary Outcome: Number of Patients With Maximum Common Toxicity Criteria - National Cancer Institute (CTC-NCI): Possibly Related to Study Drug by Grade
Description: Grades range from 0 (no toxicity) to 4 (life-threatening or disabling).
Time Frame: every 21 day cycle (6-8 cycles) and every 3 months during long-term follow-up
Measure: Number; unit: participants
Arm/Group | Gemcitabine + Cisplatin
Number analyzed (Participants) | 50
participants
  Patients with at least one CTC - Grade 1 | 34
  Patients with at least one CTC - Grade 2 | 6
  Patients with at least one CTC - Grade 3 | 2
  Patients with at least one CTC - Grade 4 | 1
  Other auditory/hearing - Grade 1 | 0
  Other auditory/hearing - Grade 2 | 0
  Other auditory/hearing - Grade 3 | 1
  Other auditory/hearing - Grade 4 | 0
  Leukocytes - Grade 1 | 0
  Leukocytes - Grade 2 | 0
  Leukocytes - Grade 3 | 0
  Leukocytes - Grade 4 | 1
  Neutrophils/granulocytes - Grade 1 | 0
  Neutrophils/granulocytes - Grade 2 | 0
  Neutrophils/granulocytes - Grade 3 | 0
  Neutrophils/granulocytes - Grade 4 | 1
  Fatigue - Grade 1 | 11
  Fatigue - Grade 2 | 0
  Fatigue - Grade 3 | 1
  Fatigue - Grade 4 | 0
  Weight loss - Grade 1 | 0
  Weight loss - Grade 2 | 1
  Weight loss - Grade 3 | 0
  Weight loss - Grade 4 | 0
  Alopecia - Grade 1 | 1
  Alopecia - Grade 2 | 1
  Alopecia - Grade 3 | 0
  Alopecia - Grade 4 | 0
  Rash/desquamation - Grade 1 | 2
  Rash/desquamation - Grade 2 | 0
  Rash/desquamation - Grade 3 | 1
  Rash/desquamation - Grade 4 | 0
  Anorexia - Grade 1 | 1
  Anorexia - Grade 2 | 0
  Anorexia - Grade 3 | 0
  Anorexia - Grade 4 | 0
  Diarrhea (without colostomy) - Grade 1 | 0
  Diarrhea (without colostomy) - Grade 2 | 0
  Diarrhea (without colostomy) - Grade 3 | 1
  Diarrhea (without colostomy) - Grade 4 | 0
  Nausea - Grade 1 | 29
  Nausea - Grade 2 | 2
  Nausea - Grade 3 | 0
  Nausea - Grade 4 | 0
  Other Gastrointestinal - Grade 1 | 0
  Other Gastrointestinal - Grade 2 | 1
  Other Gastrointestinal - Grade 3 | 0
  Other Gastrointestinal - Grade 4 | 0
  Stomatitis/pharyngitis - Grade 1 | 0
  Stomatitis/pharyngitis - Grade 2 | 0
  Stomatitis/pharyngitis - Grade 3 | 1
  Stomatitis/pharyngitis - Grade 4 | 0
  Vomiting - Grade 1 | 24
  Vomiting - Grade 2 | 0
  Vomiting - Grade 3 | 0
  Vomiting - Grade 4 | 0
  Alkaline phosphatase - Grade 1 | 13
  Alkaline phosphatase - Grade 2 | 1
  Alkaline phosphatase - Grade 3 | 0
  Alkaline phosphatase - Grade 4 | 0
  Bilirubin - Grade 1 | 6
  Bilirubin - Grade 2 | 0
  Bilirubin - Grade 3 | 0
  Bilirubin - Grade 4 | 0
  Serum glutamic oxaloacetic transaminase - Grade 1 | 8
  Serum glutamic oxaloacetic transaminase - Grade 2 | 0
  Serum glutamic oxaloacetic transaminase - Grade 3 | 0
  Serum glutamic oxaloacetic transaminase - Grade 4 | 0
  Serum glutamic pyruvic transaminase - Grade 1 | 7
  Serum glutamic pyruvic transaminase - Grade 2 | 0
  Serum glutamic pyruvic transaminase - Grade 3 | 0
  Serum glutamic pyruvic transaminase - Grade 4 | 0
  Dizziness/lightheadedness - Grade 1 | 1
  Dizziness/lightheadedness - Grade 2 | 0
  Dizziness/lightheadedness - Grade 3 | 0
  Dizziness/lightheadedness - Grade 4 | 0
  Headache - Grade 1 | 0
  Headache - Grade 2 | 1
  Headache - Grade 3 | 0
  Headache - Grade 4 | 0
  Creatinine - Grade 1 | 7
  Creatinine - Grade 2 | 1
  Creatinine - Grade 3 | 0
  Creatinine - Grade 4 | 0
  Renal failure - Grade 1 | 0
  Renal failure - Grade 2 | 0
  Renal failure - Grade 3 | 1
  Renal failure - Grade 4 | 0
  Renal/genitourinary - Other - Grade 1 | 6
  Renal/genitourinary - Other - Grade 2 | 2
  Renal/genitourinary - Other - Grade 3 | 1
  Renal/genitourinary - Other - Grade 4 | 0

ADVERSE EVENTS:
Arm/Group | Gemcitabine + Cisplatin
Serious Adverse Events (participants affected / at risk) | 2
Other Adverse Events (participants affected / at risk) | 48
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Gemcitabine + Cisplatin
Leukopenia (Blood and lymphatic system disorders) | 1/50 (1)
Neutropenia (Blood and lymphatic system disorders) | 1/50 (1)
Deafness (Ear and labyrinth disorders) | 1/50 (1)
Renal failure acute (Renal and urinary disorders) | 1/50 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk (number of events):
Term (organ system) | Gemcitabine + Cisplatin
Nausea (Gastrointestinal disorders) | 32/50 (42)
Vomiting (Gastrointestinal disorders) | 25/50 (29)
Asthenia (General disorders) | 17/50 (19)
Respiratory tract infection viral (Infections and infestations) | 4/50 (4)
Alanine aminotransferase increased (Investigations) | 9/50 (14)
Aspartate aminotransferase increased (Investigations) | 14/50 (16)
Blood alkaline phosphatase increased (Investigations) | 15/50 (15)
Blood bilirubin increased (Investigations) | 8/50 (9)
Blood creatinine increased (Investigations) | 10/50 (17)
Creatinine renal clearance decreased (Investigations) | 9/50 (12)
Weight decreased (Investigations) | 11/50 (11)
Weight increased (Investigations) | 9/50 (9)
Rash (Skin and subcutaneous tissue disorders) | 3/50 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days